CLINICAL TRIAL: NCT02054494
Title: Myocardial T1-mapping and T1-derived Extracellular Volume Fraction (ECV) in HIV-infection Patients With Chronic High and Low CD4+ Counts and in a Healthy Control Group
Brief Title: T1 Mapping in HIV Patients With High and Low CD4+ Cell Counts
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Claas P. Naehle, PD Dr. med., University Hospital, Bonn
Other Study IDs: 038/13
Record Dates: First submitted 2014-01-31; First posted 2014-02-04 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Heart Diseases; HIV
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- HIV patients with high CD4+ cell counts: HIV Infection, Chronic high CD4+ cell counts (>500 /μl), No known cardiac disease
- HIV patients with low CD4+ cell counts: HIV Infection, Chronic low CD4+ cell counts (<200 /μl), No known cardiac disease
- Control Group: No known cardiac disease.

SUMMARY:
HIV-infection is associated with an increased risk for cardiovascular disease. Especially patients with low CD4+ counts have a higher incidence of structural heart disease. Myocardial T1 relaxation time, as well as T1-derived extracellular volume fraction are relatively new methods for non-invasive myocardial tissue characterization, including diffuse myocardial fibrosis.

In our study HIV-patients with high and low CD4+ counts are examined on a 3T MRI scanner (Ingenia 3T, Philips Medical, Best, Netherlands). Scanning protocol includes common SSFP sequences, STIR imaging and LGE [Late gadolinium enhancement]. All HIV patients are treated in the HIV outpatient clinic of the hospital's Internal Medicine department and have an unremarkable history of cardiac disease. Patients are recruited from all over Germany. In order to obtain reference values, a subgroup of healthy, age-matched controls is included in this study.

Aim of this study is to show differences in T1- and ECV-values in the investigated subgroups. In addition, we also want to create cut-off values for healthy and affected myocardium in asymptomatic HIV-infected patients. This study could show whether myocardial T1 mapping is a potential screening parameter for beginning heart disease as part of an HIV-infection, and whether an application in routine diagnostic is reasonable.

ELIGIBILITY:
Inclusion Criteria:

* chronic HIV infection
* no known cardiac disease
* no cardiovascular risk factors

Exclusion Criteria:

* contraindications to MRI (e.g. metal implants)
* chronic kidney disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV patients are recruted from the HIV outpatients clinic of our hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Native T1 Relaxation Times | Measurement will be performed within 2 weeks after MRI scan
  T1 relaxation times will be directly obtained form the T1 maps through ROI analysis. T1 maps will be analyzed using a segmental approach. T1 relaxation times are given in [ms].

SECONDARY OUTCOMES:
Extracellular volume fraction (ECV) | Measurement will be performed within 2 weeks after MRI scan
  Hematocrit corrected ECV will be calculated using pre- and post-contrast T1 values for myocardium and blood pool using following formula:
  ECV= (1⁄T1 "myocardium post contrast"-1⁄T1 "myocadium pre contrast")/(1⁄T1 "blood post contrast"-1⁄ T1 "blood pre contrast") x (1-hematocrit).
  ECV is given in percentage.

OTHER OUTCOMES:
Cardiac function and aortic distensibility | Measurement will be performed within 2 weeks after MRI scan
  Cardiac function (left ventricular endsystolic volume (LV-ESV), left ventricular enddiastolic volume (LV-EDV), and left ventricular ejection fraction (LV-EF)) will be determined offline using a dedicated software (ViewForum, Philips Healthcare, Best, The Netherlands). LV-ESV and LV-EDV will be quantified manually by tracing the endocardial borders. LV-EF is given in percentage. LV-ESV and LV-EDV are given in [ml].
  Aortic Distensibility will be calculated as:
  Distensibility(10^-3 mmHg^-1 )=(Amax-Amin)/Amin x (Sys-Dias),where Amax and Amin represent the maximal and minimal cross-sectional area of the aorta on cine CMR images, and Sys and Dias represent the systolic and diastolic blood pressures (in millimetres of mercury), respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Claas P Naehle, MD, Principal Investigator — University of Bonn, Dept. of Radiology, Sigmund-Freud-Str. 25, 53127 Bonn, Germany
Locations (1):
- University of Bonn, Dept. of Radiology, Bonn, North Rhine-Westphalia, Germany